CLINICAL TRIAL: NCT00971594
Title: Age, Lifestyle, Muscle Mechanisms in Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Alice S. Ryan, PhD, University of Maryland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AG0120; K01AG021457 (NIH)
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Obesity; Glucose Intolerance; Exercise Capacity
Keywords: weight loss; glucose metabolism
MeSH Terms: conditions — Obesity; Glucose Intolerance; Weight Loss | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WL+AEX (Experimental): Weight loss plus aerobic exercise
  Interventions: Behavioral: Dietary counseling; Behavioral: AEX

INTERVENTIONS:
Behavioral: Dietary counseling — 1 hour sessions, once per week, with a registered dietitian on the American Heart Association Step I diet with caloric intake for each volunteer adjusted by the dietitian to elicit a WL of ~0.2-0.4 kg/wk
Behavioral: AEX — Moderate aerobic exercise (75-80% HRR for 45 min) at the Baltimore GRECC exercise facility using treadmills 3 times per week for 6 months.

SUMMARY:
The purpose of this study is to investigate the mechanisms by which physical inactivity and obesity alter skeletal muscle insulin signaling to cause insulin resistance and increase the development of impaired glucose tolerance (IGT).

DETAILED DESCRIPTION:
Aging is associated with a progressive development of impaired glucose tolerance (IGT), due to an increased peripheral tissue resistance to the action of insulin. Insulin resistance, a common state in both obese and sedentary individuals, eventually leads to the development of glucose intolerance, and type 2 diabetes with aging. Even in the absence of diabetes, insulin resistance is a key feature in various metabolic abnormalities that increase the risk for developing cardiovascular disease (CVD). Previous studies demonstrate improvements in glucose tolerance and glucose utilization following moderate energy restriction coupled with moderate intensity AEX. WL, through behavioral modification of diet and aerobic exercise (AEX), is perhaps the most effective way to treat as well as prevent insulin resistance and its associated metabolic complications of IGT and type 2 diabetes. Although these studies demonstrate the beneficial effect of weight loss (WL) and AEX on glucose tolerance and insulin action, not much is known about the cellular and molecular mechanisms by which these nonpharmacologic treatments improve glucose utilization in high-risk obese older individuals.

This study seeks to determine the cellular mechanisms by which aerobic exercise and weight loss alter skeletal muscle insulin signaling to improve insulin action in older glucose intolerant individuals. A second purpose is to determine whether certain genes (hereditary information) affect the way the body utilizes glucose in response to exercise and weight loss. In addition, adipose tissue is increasingly recognized as more than an inert depot serving not only to accept and store excess energy in the form of triglycerides, but also to secrete hormones and adipokines that have substantial effects on lipid and glucose metabolism. Furthermore, there are depot differences in metabolic function, as well as adipokine content. However, the physiology both underlying and consequential to these observations remains unknown. Thus, a third aim is to examine the effects of obesity on regional adipokine secretion and expression, and the relationship of adipokines to insulin resistance and the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Men older than 50 yrs of age
* Non-smoking (more than 5 years)
* BMI greater than 25 kg/m2 and less than 50 kg/m2

Exclusion Criteria:

* CAD, CHF, Myocardial infarction within 6 months or other symptomatic heart disease
* History of stroke, peripheral arterial disease
* Currently being treated for active cancer
* On oral agents or insulin therapy for diabetes
* Poorly controlled Dyslipidemia (abnormal concentration of lipids or lipoproteins in the blood)
* Poorly controlled hypertension (BP > 180/95)
* Other systematic disorders that are not medically treated and stable
* Physical impairment limiting normal activity and other contraindications to exercise
* Aerobically conditioned
* Abnormal response to exercise (chest pain, significant arrhythmias, extreme shortness of breath, cyanosis, exercising BP > 240/120)
* Taking warfarin/coumadin
* Taking oral steroids
* Abnormal renal function or liver function
* Chronic pulmonary disease severe enough to require oxygen
* Anemia
* MMSE < 24, dementia

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Insulin stimulated glucose disposal | Baseline and 6 months
Content and activity of insulin signaling proteins from muscle biopsies | Baseline and 6 months
Glucose tolerance | Baseline and 6 months

SECONDARY OUTCOMES:
Aerobic capacity | Baseline and 6 months
Body weight/Composition | Baseline and 6 months
Cytokines | Baseline and 6 months
Other biomarkers (such as glucose, insulin etc) | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Joseph, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (2):
- United States (2):
  - Baltimore VA Medical Center, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Houmard JA, Tanner CJ, Slentz CA, Duscha BD, McCartney JS, Kraus WE. Effect of the volume and intensity of exercise training on insulin sensitivity. J Appl Physiol (1985). 2004 Jan;96(1):101-6. doi: 10.1152/japplphysiol.00707.2003. Epub 2003 Sep 12. PMID 12972442
- [Background] Deshmukh AS, Hawley JA, Zierath JR. Exercise-induced phospho-proteins in skeletal muscle. Int J Obes (Lond). 2008 Sep;32 Suppl 4:S18-23. doi: 10.1038/ijo.2008.118. PMID 18719593
- [Background] Catenacci VA, Hill JO, Wyatt HR. The obesity epidemic. Clin Chest Med. 2009 Sep;30(3):415-44, vii. doi: 10.1016/j.ccm.2009.05.001. PMID 19700042
- [Derived] Prior SJ, Blumenthal JB, Katzel LI, Goldberg AP, Ryan AS. Increased skeletal muscle capillarization after aerobic exercise training and weight loss improves insulin sensitivity in adults with IGT. Diabetes Care. 2014 May;37(5):1469-75. doi: 10.2337/dc13-2358. Epub 2014 Mar 4. PMID 24595633